CLINICAL TRIAL: NCT00794547
Title: A Phase I/II Clinical Trial of Intravenous (IV) Calcitriol With Fixed Dose of Cisplatin and Docetaxel in Advanced Non-Small Cell Lung Cancer
Brief Title: Phase I/II Calcitriol in Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2008.042; HUM 21242 (Other: University of Michigan Medical IRB); NCT00470431 (obsolete NCT alias)
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: lung cancer; nsclc
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): In the Phase I part of the study, we will test the safety of calcitriol along with standard chemotherapy. In addition, the goal is to see what effects (good and bad) it has on you and your type of Non-Small Cell Lung Cancer. This study is ongoing. In this portion of the study, we are testing increasing doses of calcitriol in combination with standard chemotherapy. If 2/3 patients at any dose level experience side effects that are limiting, we will call the dose level below that dose the maximum tolerated dose.
  Interventions: Drug: Calcitriol
- 2 (Experimental): In the Phase II part of the study, we will find out the response of subjects' cancer has to the combination of a fixed dose of calcitriol (determined in the phase I study) with standard chemotherapy.
  Interventions: Drug: Calcitriol

INTERVENTIONS:
Drug: Calcitriol — Escalating dose of Calcitriol will be infused IV over 1 hour every 21 days.
  Arms: 1
Drug: Calcitriol — In this portion of the study, all patients will get the same dose of calcitriol (determined from the Phase I study) along with the standard chemotherapy
  Arms: 2

SUMMARY:
According to the Cancer Atlas, lung cancer remains the major cancer among the 10.9 million new cases of cancer diagnosed annually worldwide. The mortality from lung cancer is greater than the combined mortality for breast, colon and prostate cancer combined. Most patients with metastatic non-small-cell lung cancer (NSCLC) are treated with platinum-based chemotherapy regimens. The drug combination of cisplatin and docetaxel is one of the commonly used regimens in metastatic NSCLC. Although both drugs are powerful disruptors of cell growth, positive therapeutic response rates to this therapy remain low for NSCLC patients, from 25% to 30%. While adding new biologics such as bevacizumab to the current treatment standard can improve treatment response, median survival for advanced NSCLC patients receiving this type of treatment remains low at under 12 months. Research studies have demonstrated that Vitamin D, and it's signaling pathways are important biological targets in cancer therapeutics. In vitro and in vivo calcitriol (1, 25 dihydroxycholecalciferol) is antiproliferative and potentiates the antitumor effects of cytotoxic agents (e.g. taxanes, platinum analogues). We have shown that administration of high doses of calcitriol and cisplatin is feasible and associated with complete tumor regressions in dogs with spontaneous cancers. Calcitriol has also shown to be synergistic with docetaxel both in preclinical as well as in a recent phase II clinical trial in prostate cancer. Based on these results and other supporting data from studies indicating that calcitriol functions as a potent and well tolerated anti-tumor agent when used in combination with drugs likes cisplatin and docetaxel, we hypothesize that introducing calcitriol into treatment regimes for NSCLC patients has the potential to demonstrably improve treatment response for these patients. The overall goals for conducting this phase I/II clinical study will be (1) to determine the maximum tolerated dose (MTD) and dose limiting toxicities (DLT) of calcitriol in combination with cisplatin/docetaxel in patients with advanced NSCLC, (2) to assess the response rates of patients with advanced NSCLC to the combination of calcitriol with cisplatin/docetaxel, (3) to evaluate the pharmacokinetics (PK) of administering calcitriol intravenously at the MTD, and (4) to evaluate correlations between calcitriol PK and changes on specific coding regions of the gene associated with calcitriol breakdown.

ELIGIBILITY:
Inclusion Criteria:

1. Proven histological or cytological diagnosis of stage IIIB (malignant pleural effusion) IV NSCLC.
2. Age more than 18 years
3. Performance status must be ECOG 0-1.
4. No prior or concurrent malignancy, except non-melanoma skin cancer, or CIS of the cervix, unless documented disease-free for more than 2 years.
5. No prior use of chemotherapy for stage IV NSCLC; Adjuvant therapy is permitted.
6. Adequate bone marrow, hepatic, and renal function, as evidenced by the following: WBC 3.0 x 109/L, neutrophils 1.5 x 109 /L; platelet count 100 x 109/L; Hgb> 10 g/dL (may be transfused to 10g/dL); total bilirubin within the upper limit of the institutional normal range; (transaminases SGOT or SGPT) 1.5 times the upper limit of the institutional normal range. Creatinine within the upper limit of the institutional normal range; creatinine clearance >50 ml/min
7. Patients must have measurable or evaluable disease (not required for the phase I part of the study)
8. Normal cardiac function with no history of uncontrolled heart disease
9. Female patients must not be pregnant; they must be post-menopausal or practicing an accepted form of birth control. If pregnancy is a possibility, a pregnancy test will be required prior to initiation of therapy.
10. Life expectancy of at least 12 weeks.
11. Patient and investigator signed study-specific consent form, indicating the investigational nature of the study
12. Patients must be accessible for treatment and follow-up.
13. No chemotherapy or radiotherapy within 3 weeks of study entry defined here as day 1 of therapy with calcitriol plus chemotherapy (6 weeks for mitomycin C or a nitrosourea).
14. No treatment with investigational drugs within 3 weeks of study entry.
15. No other serious illness or medical condition including unstable cardiac disease requiring treatment, new onset crescendo or rest angina; history of significant neurological or psychiatric disorders including psychotic disorders, dementia, or seizures; or active infection are permitted. No evidence of grade > 2 peripheral neuropathy. No history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
16. Palliative radiation is permitted (as long as marrow exposed not greater than 10%; please see Appendix IV for reference) At least 1 week since the last palliative XRT.
17. Treated brain metastasis allowed with no waiting period following gamma knife and at least 2 weeks after whole brain XRT as long as neurologically stable.

Exclusion Criteria:

1. Known hypersensitivity to Vitamin D, docetaxel, cisplatin
2. Hypercalcemia (patients with serum albumin corrected calcium* > 10.7 mg/dL)
3. History of renal/bladder stones over the past 10 years
4. History of nephrectomy.
5. Uncontrolled heart disease, unstable angina, heart failure, current digoxin therapy
6. Thiazide, Digoxin or glucocorticoid therapy (except the pre-medication Dexamethasone used in the study as prescribed)
7. Unwillingness to stop calcium supplementation
8. Concurrent use of Phenytoin, Barbiturates, Rifampin, Carbamazepine, Phenobarbital or St John's wort.
9. Treatment with any investigational drug within 3 weeks before Day 1 of protocol
10. Any unresolved toxicity (NCI CTCAE version 3.0,>2) (Please see appendix V for link)
11. Pregnancy/Lactation
12. Patients with IIIB NSCLC who are eligible for definitive chemoradiation.

    * Ca corrected = Ca (measured) + (0.8 x (4 - albumin))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-12; Primary Completion 2011-10 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nithya Ramnath, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (4):
- United States (4):
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York

REFERENCES:
- [Result] Ramnath N, Daignault-Newton S, Dy GK, Muindi JR, Adjei A, Elingrod VL, Kalemkerian GP, Cease KB, Stella PJ, Brenner DE, Troeschel S, Johnson CS, Trump DL. A phase I/II pharmacokinetic and pharmacogenomic study of calcitriol in combination with cisplatin and docetaxel in advanced non-small-cell lung cancer. Cancer Chemother Pharmacol. 2013 May;71(5):1173-82. doi: 10.1007/s00280-013-2109-x. Epub 2013 Feb 23. PMID 23435876

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: In the Phase I part of the study, we will test the safety of calcitriol along with standard chemotherapy. In addition, the goal is to see what effects (good and bad) it has on you and your type of Non-Small Cell Lung Cancer. This study is ongoing. In this portion of the study, we are testing increasing doses of calcitriol in combination with standard chemotherapy. If 2/3 patients at any dose level experience side effects that are limiting, we will call the dose level below that dose the maximum tolerated dose.
  Calcitriol: Escalating dose of Calcitriol will be infused IV over 1 hour every 21 days.
- Phase 2: In the Phase II part of the study, we will find out the response of subjects' cancer has to the combination of a fixed dose of calcitriol (determined in the phase I study) with standard chemotherapy.
  Calcitriol: In this portion of the study, all patients will get the same dose of calcitriol (determined from the Phase I study) along with the standard chemotherapy
Period: Overall Study
Arm/Group | Phase 1 | Phase 2
Started | 18 | 16
Completed | 18 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Thirty-four patients were enrolled (18 in phase I and 16 in phase II).
Groups:
- Calcitriol + Cisplatin + Docetaxel: Calcitriol, administered IV at 30, 45, 60, 80, or 100 mcg/m^2 (every 21 days), along with Cisplatin, 75 mg/m^2 (every three weeks), and Docetaxel, 75 mg/m^2 (every three weeks).
Arm/Group | Calcitriol + Cisplatin + Docetaxel
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 54 [34 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 34
Histology [Number; unit: participants] — Tumor histology results. Categories include Adenocarcinoma, Squamous Carcinoma and Non-Small-Cell Lung Cancer Not Otherwise Specified (NSCLC NOS).
  participants
    Adenocarcinoma | 21
    Squamous carcinoma | 12
    NSCLC NOS | 1
Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group Performance Status at baseline. Scores may be 0 (Asymptomatic; fully active, able to carry on all predisease activities without restriction) or 1 (Symptomatic but completely ambulatory; restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. For example, light housework, office work)
  participants
    Performance Status 0 | 16
    Performance Status 1 | 18
Smoking Status [Number; unit: participants]
  Never Smoker | 2
  Ever Smoker | 29
  Unknown | 3

OUTCOME MEASURES:

1. Primary Outcome: MTD of Intravenous Calcitriol When Administered Prior to Fixed Dose Cisplatin 75mg/m2 and Docetaxel 75 mg/m2, Every 3 Weeks in Patients With Advanced Non-small Cell Lung Cancer (NSCLC)
Description: The primary objective was to determine the Maximum Tolerated Dose (MTD) of intravenous calcitriol when administered prior to fixed dose cisplatin 75mg/m2 and docetaxel 75 mg/m2, every 3 weeks in patients with advanced non-small cell lung cancer (NSCLC). Accrual duration for the study is 5 years.
Time Frame: 5 years
Population: Eighteen patients were enrolled, and 16 were evaluable for toxicity assessments. Two patients were not evaluable as they progressed prior to completion of cycle 1.
Measure: Number; unit: mcg/m^2
Arm/Group | Calcitriol + Cisplatin + Docetaxel
Number analyzed (Participants) | 16
mcg/m^2 | 60

2. Primary Outcome: Number of Participants That Experience Grade 3 or Greater Neutropenia
Description: The second primary objective was to characterize the toxicity and response of patients treated with a combination of calcitriol, cisplatin and docetaxel. Toxicity was assessed, in part, by noting the number of participants that experience grade 3 or greater neutropenia in each phase of the trial. Toxicities were recorded using NCI CTCAE (Common Terminology Criteria for Adverse Events) version 3.0 and were followed for 30 days after the date of withdrawal from study drug.
Time Frame: 30 days after last dose
Population: Thirty-four patients were enrolled (18 in phase I and 16 in phase II). 16 of 18 patients enrolled in the Phase 1 portion of the study were evaluable for toxicity. One patient in the phase II study went to another therapy prior to the 30 day window for a confirmatory scan and was thus excluded from analysis.
Measure: Number; unit: participants
Arm/Group | Calcitriol + Cisplatin + Docetaxel
Number analyzed (Participants) | 31
participants
  # of Phase 1 Participants w/ Grade 3+ Neutropenia | 8
  # of Phase 2 Participants w/ Grade 3+ Neutropenia | 9

3. Primary Outcome: Median Time to Progression
Description: The second primary objective was to characterize the toxicity and response of patients treated with a combination of calcitriol, cisplatin and docetaxel. To assess the response, median time to progression was determined. Progression was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 5 years
Population: 22 patients were treated at the Maximum Tolerated Dose, including 6 phase I patients who received the MTD during the phase 1 component. 1 of 6 phase 1 patients was not evaluable due to toxicity. 1 patient (of 16) in the phase 2 study went to another therapy prior to the 30 day window and was excluded from analysis. 20 patients were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Calcitriol + Cisplatin + Docetaxel
Number analyzed (Participants) | 20
months | 5.8 [3.4 to 6.5]

4. Primary Outcome: Median Overall Survival
Description: The second primary objective was to characterize the toxicity and response of patients treated with a combination of calcitriol, cisplatin and docetaxel. To assess the response, overall survival was determined.
Time Frame: 5 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Calcitriol + Cisplatin + Docetaxel
Number analyzed (Participants) | 20
months | 8.7 [7.6 to 39.4]

5. Secondary Outcome: Mean AUC 1,25-D3 Concentration at 12 and 24 Hours
Description: The mean AUC (area under the curve) concentrations of 1,25-D3 from 0-12 hours and 0-24 hours will be calculated.
Time Frame: 12 and 24 hours post dose
Population: Patients from the phase II portion of the study were included in the pharmacokinetics analysis
Measure: Mean (Standard Error); unit: h*ng/mL
Arm/Group | Calcitriol + Cisplatin + Docetaxel
Number analyzed (Participants) | 16
h*ng/mL
  AUC 0-12 Hours | 15.95 (0.92)
  AUC 0-24 Hours | 31.74 (1.92)

6. Other Pre Specified Outcome: To Correlate the Pharmacokinetic Parameters of Systemic Calcitriol Exposure (AUC) With SNPs of the 24-hydroxylase (CYP24), the Major Vitamin D3 Inactivating Enzyme.
Time Frame: 3-6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the start of study drug until 30 days after the date of withdrawal from study drug.
Arm/Group | Calcitriol + Cisplatin + Docetaxel
Serious Adverse Events (participants affected / at risk) | 20/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcitriol + Cisplatin + Docetaxel (N=34)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Low Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2 (2)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 2 (2)
Hypotension (Cardiac disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 3 (3)
Lung Infection (Infections and infestations) | 2 (2)
Upper Airway Infection (Infections and infestations) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1)
Glomerular filtration rate (Metabolism and nutrition disorders) | 1 (1)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (1)
Pain-Back (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain-Chest (Cardiac disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcitriol + Cisplatin + Docetaxel (N=34)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Tinnitus (Ear and labyrinth disorders) | 4 (5)
Low Hemoglobin (Blood and lymphatic system disorders) | 14 (23)
Low Leukocytes (total WBC) (Blood and lymphatic system disorders) | 14 (24)
Lymphopenia (Blood and lymphatic system disorders) | 11 (24)
Low Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 14 (23)
Low Platelets (Blood and lymphatic system disorders) | 8 (15)
Atrial fibrillation (Cardiac disorders) | 3 (5)
Sinus tachycardia (Cardiac disorders) | 4 (6)
Hypertension (Cardiac disorders) | 3 (3)
Hypotension (Cardiac disorders) | 7 (10)
Fatigue (General disorders) | 17 (28)
Fever (General disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (5)
Rigors/chills (General disorders) | 4 (4)
Weight loss (Investigations) | 4 (7)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 5 (5)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 7 (7)
Anorexia (Gastrointestinal disorders) | 15 (17)
Constipation (Gastrointestinal disorders) | 7 (7)
Dehydration (Gastrointestinal disorders) | 6 (10)
Diarrhea (Gastrointestinal disorders) | 10 (15)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 3 (4)
Mucositis/stomatitis (Gastrointestinal disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 21 (29)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 9 (13)
Vomiting (Gastrointestinal disorders) | 12 (16)
Febrile neutropenia (Infections and infestations) | 4 (4)
Edema: limb (General disorders) | 4 (7)
Elevated ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 5 (15)
Elevated AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 9 (13)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 11 (15)
Elevated Alkaline phosphatase (Metabolism and nutrition disorders) | 7 (12)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 4 (5)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 7 (11)
Elevated Creatinine (Metabolism and nutrition disorders) | 4 (6)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 17 (42)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 4 (6)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 6 (6)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 6 (8)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 14 (20)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (6)
Dizziness (Nervous system disorders) | 7 (8)
Neuropathy: sensory (Nervous system disorders) | 4 (5)
Vision-blurred vision (Eye disorders) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 6 (10)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (10)
Bone Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Chest Pain (Cardiac disorders) | 3 (4)
Limb Pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Head Pain (Nervous system disorders) | 5 (6)
Pain NOS (General disorders) | 3 (3)
Throat Pain (Gastrointestinal disorders) | 5 (5)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (14)
Urinary retention (Renal and urinary disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No